CLINICAL TRIAL: NCT02431689
Title: Antagonist and Short Protocols in Invitro Fertilization/Intracytoplasmic Sperm Injection (IVF/ICSI) Cycles With Delayed Embryo Transfer in Poor Ovarian Response
Brief Title: Delayed Embryo Transfer in Poor Responders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Nile Ivf Center, Cairo, Egypt (Other); Kamal Shaeer center of infertility (Unknown)
Responsible Party: Principal Investigator, Yasmin Ahmed Bassiouny, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32015
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Antagonist (Active Comparator): Antagonist protocol (fixed) for IVF/ICSI, with starting dose of human menopausal gonadotrophins (HMG) from 300-450 IU from day 1 of the cycle, antagonist start from day 6 stimulation. Follow-up by ultrasound and serum estradiol will be done. Triggering of ovulation using human chorionic gonadotrophin (HCG) 10000 IU I.M. when at least 2-3 follicles reach 17mm in diameter.
  Cryopreservation of all embryos at will be done. Frozen embryo transfer in the following cycle will be attempted using estradiol valerate (6mg) for endometrial preparation after pituitary down regulation using long acting GnRH analogue . A maximum of 3 good quality embryos will be transferred.
  Interventions: Procedure: IVF/ICSI
- Short (Active Comparator): Short protocol for IVF/ICSI, gonadotrophin releasing hormone analogue (GnRHa) starts from day 1 of the cycle, HMG starts in a dose from 300-450 IU from day 3, Follow-up by ultrasound and serum estradiol will be done. Triggering of ovulation using human chorionic gonadotrophin (HCG) 10000 IU I.M. when at least 2-3 follicles reach 17mm in diameter.
  Cryopreservation of all embryos at will be done. Frozen embryo transfer in the following cycle will be attempted using estradiol valerate (6mg) for endometrial preparation after pituitary down regulation using long acting GnRH analogue . A maximum of 3 good quality embryos will be transferred.
  Interventions: Procedure: IVF/ICSI

INTERVENTIONS:
Procedure: IVF/ICSI — controlled ovarian hyperstimulation with various protocols, follow up till stimulated follicles measure from 18-20 mm, then ovum pickup followed by embryo transfer is done.

SUMMARY:
Poor ovarian response indicates inadequate ovarian response to ovarian stimulation. In the current study the investigators will attempt to compare antagonist and short protocols regarding oocyte as well as embryo quantity and quality. Frozen embryo transfer will be performed in order to abolish iatrogenic effect of stimulation drugs on implantation. Still implantation and pregnancy rates are considered secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient selection is based on the ESHRE consensus group 2011 definition of poor ovarian response (POR) (Bologna criteria):
* At least two of the following three features must be present:

  1. Advanced maternal age (≥40 years) or any other risk factor for POR;
  2. A previous POR (≤3 oocytes with a conventional stimulation protocol);
  3. An abnormal ovarian reserve test (i.e. Antral follicle count (AFC) <5-7 follicles or Antimullerian hormone (AMH) <0.5-1.1 ng/ml).

Two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal Ovarian reserve test (ORT). By definition, the term POR refers to the ovarian response and, therefore, one stimulated cycle is considered essential for the diagnosis of POR. However, patients over 40 years of age with an abnormal ORT may be classified as poor responders since both advanced age and an abnormal ORT may indicate reduced ovarian reserve and act as a surrogate of ovarian stimulation cycle. In this case, the patients should be more properly defined as expected PORs.

Exclusion Criteria:

* Women with endometriosis, endocrinal problems, uterine abnormalities as well as male azospermia.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Number of Metaphase II (MII) oocytes | 9-14 days from stimulation
  Number of MII oocytes collected from each patient on the day of ovum pickup (OPU)
Number of good embryos | 3-5 days after ovum pickup
  the number of good quality embryos obtained from each patient

SECONDARY OUTCOMES:
chemical pregnancy rate | 14 days after embryo transfer
  positive serum Beta HCG 14 days after embryo transfer
clinical pregnancy rate | 5 weeks after embryo transfer
  the detection of intrauterine gestational sac with positive pulsations
Implantation rate | 5 weeks after embryo transfer
  the ratio between the number of embryos transferred and the number of sacs
Early miscarriage rate | 3 months
  Pregnancy loss in the first 12 weeks gestation
Ongoing pregnancy rate | 3 months
  Pregnancy ongoing beyond 12 weeks gestation
Live birth rate | 9 months
  Pregnancy ending with a live birth

CONTACTS AND LOCATIONS:
Overall Officials: Iman K Shaeer, MD, Study Director — Cairo University
Locations (3):
- Egypt (3):
  - IVF centre, Obstetrics and Gynaecology Department, Cairo University Hospitals (Kasr EL Aini), Cairo
  - Kamal Shaeer center of infertility, Giza
  - Nile IVF center, Giza

IPD SHARING:
Plan to Share IPD: No